CLINICAL TRIAL: NCT04571385
Title: A Double-Blind, Randomised, Placebo-Controlled, Parallel-Group Study of AP30663 Given Intravenously for Cardioversion in Patients With Atrial Fibrillation
Brief Title: A Study Evaluating the Efficacy and Safety of AP30663 for Cardioversion in Participants With Atrial Fibrillation (AF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acesion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP30663-2001; 2018-004445-17 (EudraCT Number)
Record Dates: First submitted 2020-09-25; First posted 2020-10-01 (Actual); Results first posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1: AP30663 (Experimental): Participants will receive single dose of AP30663.
  Interventions: Drug: AP30663
- Part 1: Placebo (Placebo Comparator): Participants will receive placebo matched to AP30663.
  Interventions: Drug: Placebo
- Part 2: AP30663 (Experimental): Participants will receive a single dose of one of the multiple dose levels of AP30663.
  Interventions: Drug: AP30663
- Part 2: Placebo (Placebo Comparator): Participants will receive placebo matched to AP30663.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AP30663 — Administer by intravenous infusion.
  Arms: Part 1: AP30663; Part 2: AP30663
Drug: Placebo — Placebo matched to AP30663.
  Arms: Part 1: Placebo; Part 2: Placebo

SUMMARY:
This study will evaluate the efficacy, safety, tolerability and pharmacokinetics (PK) of one or more doses of AP30663 for cardioversion in adult participants with AF.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical indication for cardioversion of AF
* Current episode of symptomatic AF lasting between 3-hour and 7 days (inclusive) at randomization
* Adequate anticoagulation according to international and/or national guidelines

Key Exclusion Criteria:

* Significant clinical illness or surgical procedure within 4 weeks preceding the screening visit
* History of significant mental, renal or hepatic disorder, chronic obstructive pulmonary disease, sinus nodal disease, or other significant disease, as judged by the investigator.
* Any cardioversion attempt of AF or atrial flutter within 4 weeks preceding randomization
* Use of any antiarrhythmic drug class I and/or III within 6 months before randomisation

Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2023-01-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- Denmark (5):
  - Acesion Pharma Investigational Site 110, Aalborg
  - Acesion Pharma Investigational Site 106, Copenhagen
  - Acesion Pharma Investigational Site 108, Hellerup
  - Acesion Pharma Investigational Site 113, Hillerød
  - Acesion Pharma Investigational Site 105, Roskilde
- Hungary (10):
  - Acesion Pharma Investigational Site 202, Budapest
  - Acesion Pharma Investigational Site 203, Budapest
  - Acesion Pharma Investigational Site 207, Budapest
  - Acesion Pharma Investigational Site 212, Budapest
  - Acesion Pharma Investigational Site 213, Budapest
  - Acesion Pharma Investigational Site 214, Budapest
  - Acesion Pharma Investigational Site 211, Pécs
  - Acesion Pharma Investigational Site 201, Szekszárd
  - Acesion Pharma Investigational Site 210, Szentes
  - Acesion Pharma Investigational Site 204, Zalaegerszeg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holst AG, Tomcsanyi J, Vestbjerg B, Grunnet M, Sorensen US, Diness JG, Bentzen BH, Edvardsson N, Hohnloser SH, Bhatt DL, Dorian P. Inhibition of the KCa2 potassium channel in atrial fibrillation: a randomized phase 2 trial. Nat Med. 2024 Jan;30(1):106-111. doi: 10.1038/s41591-023-02679-9. Epub 2023 Dec 13. PMID 38092897

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 8 active sites in 2 countries (Denmark and Hungary) from 09 September 2019 to 23 January 2023.
Pre-assignment Details: A total of 66 participants were enrolled, of which 63 participants received the study treatment in 2 parts. Part 1 consists of Placebo and AP30663 (3 milligrams per kilogram [mg/kg]) and part 2 consist of Placebo and AP30663 (5 mg/kg). As per the planned statistical analysis, placebo arms with similar dosing strategies in Part 1 and Part 2 were combined to be reported as a pooled placebo arm.
Groups:
- Part 1 and 2: Pooled Placebo: Participants received a single intravenous (IV) infusion of AP30663 matched placebo for 30 minutes on Day 1 in both Part 1 and 2.
- Part 1: AP30663 3mg/kg: Participants received a single IV infusion of AP30663 3mg/kg for 30 minutes on Day 1 in Part 1.
- Part 2: AP30663 5mg/kg: Participants received a single IV infusion of AP30663 5mg/kg for 30 minutes on Day 1 in Part 2.
Period: Overall Study
Arm/Group | Part 1 and 2: Pooled Placebo | Part 1: AP30663 3mg/kg | Part 2: AP30663 5mg/kg
Started | 27 | 16 | 23
Part 1 | 16 | 16 | 0
Part 2 | 11 | 0 | 23
Full Analysis Set (FAS) (Full Analysis Set included all randomized participants who were administered double-blind study treatment and had an evaluable Atrial Fibrillation conversion status within 90 minutes from the start of infusion.) | 25 | 12 | 22
Safety Set (Safety set included all randomized participants who were administered double-blind study treatment and had analyzed according to the treatment received.) | 26 | 15 | 22
Pharmacokinetic (PK) Set (The Pharmacokinetic Set included all participants in the Safety Set who had at least one evaluable post-baseline drug concentration value.) | 0 | 15 | 22
Treated | 26 | 15 | 22
Completed | 26 | 15 | 22
Not Completed | 1 | 1 | 1
Not completed — Participant non-compliance | 1 | 0 | 0
Not completed — Converted to Sinus Rhythm (SR) before the infusion | 0 | 1 | 0
Not completed — Screen failure | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety set included all randomized participants who were administered double-blind study treatment and had analyzed according to the treatment received.
Groups:
- Part 1 and 2: Pooled Placebo: Participants received a single IV infusion of AP30663 matched placebo for 30 minutes on Day 1 in both Part 1 and 2.
- Total: Total of all reporting groups
Arm/Group | Part 1 and 2: Pooled Placebo | Part 1: AP30663 3mg/kg | Part 2: AP30663 5mg/kg | Total
Number analyzed (Participants) | 26 | 15 | 22 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (9.23) | 65.4 (8.48) | 65.5 (10.38) | 65.0 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 7 | 18
  Male | 18 | 12 | 15 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 15 | 22 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Converted From Atrial Fibrillation (AF) Within 90 Minutes From Start of Infusion and Subsequently Had no AF Recurrence Within 1 Minute of Conversion From AF
Description: The 12-lead Holter monitoring equipment was used to monitor heart rate and its rhythm. Electrocardiogram (ECG) was performed in a standardized manner after the participant had rested in the semi-supine position for at least 5 minutes. Conversion from AF to normal sinus rhythm within 90 minutes from start of infusion was determined by the investigator and documented with a rhythm strip confirming conversion. Percentages were based on "number of participants converted from atrial fibrillation and absence of recurrence of AF within 1 minute of conversion" divided by "total number of participants" *100 in each treatment group. Analysis was performed based on Bayesian model.
Time Frame: Within 90 minutes from the start of infusion (Day 1)
Population: Full Analysis Set included all randomized participants who were administered double-blind study treatment and had an evaluable AF conversion status within 90 minutes from the start of infusion.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1 and 2: Pooled Placebo | Part 1: AP30663 3mg/kg | Part 2: AP30663 5mg/kg
Number analyzed (Participants) | 25 | 12 | 22
Percentage of participants | 0 | 41.7 | 54.5

2. Secondary Outcome: Time to Conversion From Atrial Fibrillation From Start of Infusion
Description: The 12-lead Holter monitoring equipment was used to monitor heart rate and its rhythm. ECG was performed in a standardized manner after the participant had rested in the semi-supine position for at least 5 minutes. Time to conversion (in minutes) was calculated by time of conversion or censoring minus time of start of infusion.
Time Frame: From start of infusion (Day 1) up to Day 2
Population: Full Analysis Set included all randomized participants who were administered double-blind study treatment and had an evaluable AF conversion status within 90 minutes from the start of infusion. Here, "overall number of participants analyzed" signifies those participants were evaluable for this outcome measure. No participant had conversion from AF to normal rhythm in placebo arm.
Measure: Median (Full Range); unit: Minutes
Arm/Group | Part 1 and 2: Pooled Placebo | Part 1: AP30663 3mg/kg | Part 2: AP30663 5mg/kg
Number analyzed (Participants) | 0 | 5 | 12
Minutes |  | 42.0 [24 to 81] | 35.0 [19 to 89]

3. Secondary Outcome: Percentage of Participants With Relapse of AF Within 5 Minutes (IRAF) After Pharmacological or Direct Current (DC) Cardioversion
Description: The 12-lead Holter monitoring equipment was used to monitor heart rate and its rhythm. ECG was performed in a standardized manner after the participant had rested in the semi-supine position for at least 5 minutes. Participants with relapse of AF within 5 minutes following pharmacological or DC cardioversion was presented by treatment and analyzed using a logistic regression model. Percentages were based on "number of participants with relapse of AF within 5 minutes after Pharmacological or DC cardioversion" divided by "total number of participants" *100 in each treatment group.
Time Frame: Within 5 minutes after cardioversion (Day 1)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1 and 2: Pooled Placebo | Part 1: AP30663 3mg/kg | Part 2: AP30663 5mg/kg
Number analyzed (Participants) | 25 | 12 | 22
Percentage of participants | 4.0 | 0 | 0

4. Secondary Outcome: Percentage of Participants With Sinus Rhythm (SR) at 3 Hours, 24 Hours and Day 30 After Start of Infusion
Description: The 12-lead Holter monitoring equipment was used to monitor heart rate and its rhythm. ECG was performed in a standardized manner that the participant had rested in the semi-supine position for at least 5 minutes. Percentage of participants in SR was assessed from Holter ECGs at 3 hours, 24 hours and Day 30 after start of infusion. Percentages were based on "number of participants in SR at 3 hours, 24 hours and Day 30 after start of infusion" divided by "total number of participants" *100 in each treatment group.
Time Frame: At 3 hours, 24 hours and Day 30 after start of Infusion (Day 1)
Population: Full Analysis Set included all randomized participants who were administered double-blind study treatment and had an evaluable AF conversion status within 90 minutes from the start of infusion. Here, "overall number of participants analyzed" signifies those participants were evaluable for this outcome and "number analyzed" signifies participants at specific timepoints.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1 and 2: Pooled Placebo | Part 1: AP30663 3mg/kg | Part 2: AP30663 5mg/kg
Number analyzed (Participants) | 25 | 11 | 21
Percentage of participants
  Sinus Rhythm at 3 hours | 84.0 | 100.0 | 95.2
  Sinus Rhythm at 24 hours | 76.0 | 100.0 | 100.0
  Sinus Rhythm at Day 30: number analyzed (Participants) | 25 | 10 | 21
  Sinus Rhythm at Day 30 | 64.0 | 90.0 | 71.4

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. TEAEs are defined as any AE occurring or worsening on or after the first dose of study medication. A serious adverse event (SAE) is defined as any serious adverse event that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, significant medical events that may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed before. TEAEs include both serious and non-serious adverse events.
Time Frame: From start of infusion (Day 1) up to follow-up (Day 35)
Population: Safety set included all randomized participants who were administered double-blind study treatment. Participants analyzed according to the treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 and 2: Pooled Placebo | Part 1: AP30663 3mg/kg | Part 2: AP30663 5mg/kg
Number analyzed (Participants) | 26 | 15 | 22
Participants
  Participants with TEAEs | 13 | 4 | 11
  Participants with Serious TEAEs | 4 | 0 | 0

6. Secondary Outcome: Changes From Baseline in Fridericia's Correction of QT Interval (ΔQTcF) Interval Data Over Time
Description: QTcF was assessed based on 12-lead Holter monitoring equipment. Triplicate ECGs were extracted at the same time points as PK sampling and were read in a semi-automated manner by a blinded cardiologist. The participant rested in the semi-supine position for at least 5 minutes at ECG extraction timepoints. Change from baseline was estimated based on a linear mixed-effects model: ΔQTcF = Time + Treatment + Time*Treatment + Baseline QTcF.
Time Frame: Baseline, 15 minutes, 45 minutes, 2 hours, 8 hours and 24 hours post-dose
Population: All randomized participants who were administered double-blind study treatment and with measurements at baseline as well as on-treatment with at least 1 post-dose time point with a valid ΔQTcF value. Participants were analyzed according to the treatment received. Here, "number analyzed" signifies those participants were evaluable at specific timepoints.
Measure: Least Squares Mean (Standard Error); unit: Millisecond
Arm/Group | Part 1 and 2: Pooled Placebo | Part 1: AP30663 3mg/kg | Part 2: AP30663 5mg/kg
Number analyzed (Participants) | 26 | 15 | 22
Millisecond
  Change at 15 minutes post-dose | 1.9 (3.21) | 11.7 (4.26) | 21.2 (3.49)
  Change at 45 minutes post-dose: number analyzed (Participants) | 26 | 15 | 21
  Change at 45 minutes post-dose | 1.0 (3.21) | 19.4 (4.26) | 37.7 (3.53)
  Change at 2 hours post-dose: number analyzed (Participants) | 14 | 15 | 0
  Change at 2 hours post-dose | 6.2 (3.93) | 23.0 (4.26) |
  Change at 8 hours post-dose: number analyzed (Participants) | 24 | 14 | 20
  Change at 8 hours post-dose | 11.5 (3.29) | 13.6 (4.34) | 17.2 (3.59)
  Change at 24 hours post-dose: number analyzed (Participants) | 16 | 11 | 10
  Change at 24 hours post-dose | 10.3 (3.74) | 14.9 (4.67) | 13.1 (4.53)

7. Secondary Outcome: Maximum Observed Peak Plasma Concentration (Cmax) of AP30663
Description: Cmax was defined as the maximum observed peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve. Blood samples were collected at indicated timepoints. Pharmacokinetics (PK) was conducted using standard noncompartmental method.
Time Frame: Baseline (pre-infusion) and at 5, 15, 25, 30, 45 minutes, 1 hour, 1.5 hours, 4 hours, 8 hours and 24 hours post-infusion
Population: The PK Set included all participants in the Safety Set who had at least one evaluable post-baseline drug concentration value.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per liter
Arm/Group | Part 1: AP30663 3mg/kg | Part 2: AP30663 5mg/kg
Number analyzed (Participants) | 15 | 22
Micrograms per liter | 7606.065 (31.5) | 10281.754 (30.9)

8. Secondary Outcome: Time to Reach Peak Plasma Concentration (Tmax) of AP30663
Description: Tmax was directly determined from concentration time data. Blood samples were collected at indicated timepoints. Pharmacokinetics was conducted using standard noncompartmental method.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: AP30663 3mg/kg | Part 2: AP30663 5mg/kg
Number analyzed (Participants) | 15 | 22
Hours | 0.4170 [0.250 to 0.500] | 0.4170 [0.250 to 1.000]

9. Secondary Outcome: Terminal Half Life of (T1/2) of AP30663
Description: T1/2 was calculated as loge (2) per elimination rate constant (kel), where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Blood samples were collected at indicated timepoints. Pharmacokinetics was conducted using standard noncompartmental method.
Time Frame: as for outcome 7
Population: The PK Set included all participants in the Safety Set who had at least one evaluable post-baseline drug concentration value. Here, "overall number of participants analyzed" signifies those participants were evaluable for this outcome.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: AP30663 3mg/kg | Part 2: AP30663 5mg/kg
Number analyzed (Participants) | 14 | 22
Hours | 5.363 [2.60 to 8.39] | 5.620 [4.35 to 8.74]

10. Secondary Outcome: Area Under the Concentration Time Curve From Pre-dose Concentration up to 30 Minutes (AUC0-0.5) of AP30663
Description: AUC0-0.5 was defined as area under the concentration time curve from pre-dose concentration up to 30 minutes. Blood samples were collected at indicated timepoints. Pharmacokinetics was conducted using standard noncompartmental method.
Time Frame: Baseline (pre-infusion) and at 5, 15, 25, 30 minutes post-infusion
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per liter
Arm/Group | Part 1: AP30663 3mg/kg | Part 2: AP30663 5mg/kg
Number analyzed (Participants) | 15 | 22
Hours*micrograms per liter | 2568.175 (41.2) | 3446.078 (79.1)

11. Secondary Outcome: Area Under the Concentration Time Curve up to the Last Measurable Concentration (AUC0-t) of AP30663
Description: AUC0-t was defined as area under the concentration-time curve from time zero to time of last measurable concentration. Blood samples were collected at indicated timepoints. Pharmacokinetics was conducted using standard noncompartmental method.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per liter
Arm/Group | Part 1: AP30663 3mg/kg | Part 2: AP30663 5mg/kg
Number analyzed (Participants) | 15 | 22
Hours*micrograms per liter | 19328.384 (44.0) | 29587.109 (31.4)

12. Secondary Outcome: Area Under the Concentration-Time Curve From Pre-dose (Zero) Through Concentration to Infinity (AUC0-inf) of AP30663
Description: AUC0-inf was defined as area under the concentration time curve from pre-dose through concentration to infinity (extrapolated), calculated as AUC0-t + Ct/Kel, where Ct is the last observed non-zero concentration. Blood samples were collected at indicated timepoints. Pharmacokinetics was conducted using standard noncompartmental method.
Time Frame: as for outcome 7
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per liter
Arm/Group | Part 1: AP30663 3mg/kg | Part 2: AP30663 5mg/kg
Number analyzed (Participants) | 14 | 22
Hours*micrograms per liter | 21623.095 (43.4) | 31448.932 (33.3)

13. Secondary Outcome: Elimination Rate Constant (Kel) of AP30663
Description: Kel represents the fraction of drug eliminated per unit of time. Elimination rate constant was calculated using linear regression on the terminal portion of the log-linear concentration versus time curve. Blood samples were collected at indicated timepoints. Pharmacokinetics was conducted using standard noncompartmental method.
Time Frame: as for outcome 7
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hour
Arm/Group | Part 1: AP30663 3mg/kg | Part 2: AP30663 5mg/kg
Number analyzed (Participants) | 14 | 22
Per hour | 0.13092 (31.4) | 0.11817 (18.6)

ADVERSE EVENTS:
Time Frame: From start of infusion (Day 1) up to follow-up (Day 35)
Description: Safety set included all randomized participants who were administered double-blind study treatment and had analyzed according to the treatment received.
Arm/Group | Part 1 and 2: Pooled Placebo | Part 1: AP30663 3mg/kg | Part 2: AP30663 5mg/kg
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/15 | 0/22
Serious Adverse Events (participants affected / at risk) | 4/26 | 0/15 | 0/22
Other Adverse Events (participants affected / at risk) | 13/26 | 4/15 | 11/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 and 2: Pooled Placebo (N=26) | Part 1: AP30663 3mg/kg (N=15) | Part 2: AP30663 5mg/kg (N=22)
Atrial fibrillation (Cardiac disorders) | 4 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 and 2: Pooled Placebo (N=26) | Part 1: AP30663 3mg/kg (N=15) | Part 2: AP30663 5mg/kg (N=22)
Atrial fibrillation (Cardiac disorders) | 7 | 1 | 7
Atrial flutter (Cardiac disorders) | 1 | 0 | 3
Atrioventricular block first degree (Cardiac disorders) | 1 | 2 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1
Phlebitis (Vascular disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 2
Dizziness postural (Nervous system disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT04571385/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-20): https://cdn.clinicaltrials.gov/large-docs/85/NCT04571385/SAP_001.pdf